CLINICAL TRIAL: NCT01603849
Title: Randomized Phase II Trial of Prophylactic Cranial Irradiation in Patients With Lung Adenocarcinoma Clinical Stage IIIB and IV With High Risk of Brain Metastasis
Brief Title: Prophylactic Cranial Irradiation in Patients With Lung Adenocarcinoma With High Risk of Brain Metastasis
Acronym: PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head of Lung Cancer Clinic, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pciHighRiskINCAN
Record Dates: First submitted 2012-04-17; First posted 2012-05-23 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer
Keywords: Prophylactic Cranial Irradiation; Lung Cancer; Non Small Cell Lung Cancer; Carcinoembryonic Antigen
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Prophylactic Cranial Irradiation (Experimental): Patients will received PCI 25 Gy in 10 fractions WBRT 4 weeks after initial treatment in the absence of disease progression.
  Interventions: Radiation: Prophylactic Cranial Irradiation
- B Observation Group (No Intervention): Patients in this arm will be observed (not receiving WBRT)

INTERVENTIONS:
Radiation: Prophylactic Cranial Irradiation — Patients allocated to this arm will received treatment with whole brain radiotherapy 25 Gy in 10 fractions.
  Arms: A Prophylactic Cranial Irradiation

SUMMARY:
Lung cancer is the first cause of death among cancer patients. Non Small Cell lung cancer (NSCLS) represents about 80-85% of the cases. Of this, about 80% presents with locally advanced or metastatic disease. Important to mention the number of patients that progress or recur in central nervous system (CNS). It has been reported that patients with adenocarcinoma, who are under 60 years and with elevated carcinoembryonic antigen (CEA) are in the highest risk to develop brain metastasis. In small cell lung cancer, treatment with prophylactic cranial irradiation (PCI) is the standard of care in patients without progression after locoregional or systemic treatment because the proven benefit in overall survival (OS) and progression free survival (PFS). However, in NSCLC PCI has not been able to prove any survival benefit, only in CNS PFS, probably because there is no trial, to our knowledge, of PCI in NSCLC that include only the specific group of patients considered in high risk of developing brain metastasis.

DETAILED DESCRIPTION:
Objectives:

1. To obtain a greater PFS and CNS PFS in patients with NSCLC treated with PCI after locoregional or systemic treatment.
2. Evaluate the benefit in OS in the specific group of patients who are at increased risk of developing brain metastasis
3. Evaluate quality of life and mental function before and after treatment with PCI and compare it with patients in the observation group.

Methods: One hundred and twenty eight patients with locally advanced or metastatic (except CNS metastasis) NSCLC will be included and randomized to receive either observation or PCI 25 Gy in 10 fractions Whole Brain Radiotherapy (WBRT) once the initial treatment has been completed and progression of the disease ruled out.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven advanced NSCLC (Stage IIIB or IV) including wild-type, EGFR-mutated or ALK-rearrangements who received treatment and were without progression at the end.
* Above 18 years
* General status with a Karnofsky >80%
* Eastern Cooperative Group (ECOG) ≤2
* Negative CNS MRI at the beginning of any treatment
* Carcinoembryonic antigen > 20 pg
* Hepatic and hematic cytology test within normal range
* Adequate renal function
* Those who accepted to participate in the study and who sign the letter of informed consent.

Exclusion Criteria:

* Patients with another type of cancer
* Patients who refuse participate in the protocol
* General status with a Karnofsky <80%
* Eastern Cooperative Group (ECOG) >2
* Previous treatment with WBRT
* Previous treatment with chemotherapy
* Disease progression after initial treatment, either chemotherapy or chemoradiotherapy depending the case.
* CNS metastasis at diagnosis
* Abnormal laboratory test that interfere with chemotherapy or TKI administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of brain metastases | 24 months
  From the day of randomization to the date when brain metastasis develop if this is the case.

SECONDARY OUTCOMES:
Overall Survival | 24 months
  From the day of randomization to the date of death if this is the case
Quality of life as per QLQ-C30 | 12 months
  a QLQ questionnaire from EORTC organization (spanish version) will be performed before, during and after PCI and will be compared with the observation group questionnaires.
Mental function | 12 months
  A mini mental status examination will be performed before, during and after PCI and will be compared with the observation group questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Oscar MD Arrieta, MD, Principal Investigator — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arrieta O, Maldonado F, Turcott JG, Zatarain-Barron ZL, Barron F, Blake-Cerda M, Cabrera-Miranda LA, Cardona AF, de la Garza JG, Rosell R. Prophylactic Cranial Irradiation Reduces Brain Metastases and Improves Overall Survival in High-Risk Metastatic Non-Small Cell Lung Cancer Patients: A Randomized phase 2 Study (PRoT-BM trial). Int J Radiat Oncol Biol Phys. 2021 Aug 1;110(5):1442-1450. doi: 10.1016/j.ijrobp.2021.02.044. Epub 2021 Feb 25. PMID 33640422